CLINICAL TRIAL: NCT05022329
Title: A Multi-Centre 12 Month Parallel-Group Randomized Control Trial of BNT162b2 Versus mRNA( Messenger Ribonucleic Acid) -1273 COVID-19 Vaccine Boosters in Chronic Kidney Disease and Dialysis Patients With Poor Humoral Response Following COVID-19 ( Corona Virus Disease of 2019)Vaccination
Brief Title: COVID-19 Vaccine Boosters in Patients With CKD
Acronym: BOOST KIDNEY
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Trial participants became eligible to receive their 4th dose of the COVID-19 vaccine vaccine thus data collected from the 12 month follow-up after 3rd dose vaccine, as per current protocol, would not not be relevant to the study outcomes.
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University Health Network, Toronto (Other); Unity Health Toronto (Other); Scarborough General Hospital (Other); Providence Healthcare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3750
Record Dates: First submitted 2021-08-23; First posted 2021-08-26 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2023-05

CONDITIONS: Chronic Kidney Diseases; COVID-19
Keywords: Vaccine; CKD
MeSH Terms: conditions — Renal Insufficiency, Chronic; COVID-19 | interventions — BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Patients who received two doses Pfizer-BioNTech vaccine, Arm 1 (Experimental)
  Interventions: Biological: Pfizer-BioNTech COVID-19 Vaccine
- Patients who received two doses MODERNA vaccine, Arm 2 (Experimental)
  Interventions: Biological: Pfizer-BioNTech COVID-19 Vaccine
- Patients who received two doses Pfizer-BioNTech vaccine ,Arm 3 (Experimental)
  Interventions: Biological: MODERNA SARS-CoV-2 Vaccine
- Patients who received two doses MODERNA vaccine, Arm 4 (Experimental)
  Interventions: Biological: MODERNA SARS-CoV-2 Vaccine

INTERVENTIONS:
Biological: Pfizer-BioNTech COVID-19 Vaccine — This arm receives Pfizer-BioNTech COVID-19 Vaccine
  Other Names: BNT162b2 mRNA COVID-19 Vaccine
  Arms: Patients who received two doses MODERNA vaccine, Arm 2; Patients who received two doses Pfizer-BioNTech vaccine, Arm 1
Biological: MODERNA SARS-CoV-2 Vaccine — This arm receives MODERNA SARS-CoV-2 Vaccine
  Other Names: mRNA-1273 SARS-CoV-2 Vaccine
  Arms: Patients who received two doses MODERNA vaccine, Arm 4; Patients who received two doses Pfizer-BioNTech vaccine ,Arm 3

SUMMARY:
This study is a 12-month, four-arm parallel-group randomized control trial of Pfizer-BioNTech versus MODERNA COVID-19 (Corona Virus disease 2019)vaccine boosters in chronic kidney disease and dialysis patients with poor humoral response following COVID-19 vaccination, in collaboration with 5 dialysis centers in Ontario and British Columbia, Canada .

Patients will be randomized to MODERNA or Pfizer-BioNTech COVID-19 vaccine, they may have received either MODERNA or Pfizer-BioNTech COVID-19 vaccine for their initial two doses of vaccine, and will be stratified by their initial vaccine type (MODERNA or Pfizer-BioNTech ) prior to randomization, which will result in four study groups.

DETAILED DESCRIPTION:
MODERNA : Nucleocapsid Modified messenger RNA BioNTech: Bio-Pharma new Technology

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic Kidney Disease (CKD)stage 3b-5 defined as an eGFR( estimated glomerular filtration rate ) of less than 45ml/min/1.73m2 or less will be eligible. Stage 5 CKD will include patients receiving in-center hemodialysis, home dialysis (home hemodialysis or peritoneal dialysis), vaccinated with two doses of the COVID-19 vaccine will be eligible for a third dose to be given 2-12 months following the second dose.
* Age ≥18 at the time of study enrolment

Exclusion Criteria:

* Patients not vaccinated against COVID-19 vaccination.
* Patients who received heterologous first two doses of vaccine
* Patients with a severe allergic reaction to prior COVID-19 vaccination or any of the ingredients.
* New COVID-19 infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Scarborough Health Network, Scarborough Village, Ontario
  - University Health Network, Toronto, Ontario
  - Sunnybrook Health Science Center, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yau K, Tam P, Chan CT, Hu Q, Qi F, Abe KT, Kurtesi A, Jiang Y, Estrada-Codecido J, Brown T, Liu L, Siwakoti A, Leis JA, Levin A, Oliver MJ, Colwill K, Gingras AC, Hladunewich MA. BNT162b2 versus mRNA-1273 Third Dose COVID-19 Vaccine in Patients with CKD and Maintenance Dialysis Patients. Clin J Am Soc Nephrol. 2024 Jan 1;19(1):85-97. doi: 10.2215/CJN.0000000000000328. Epub 2023 Oct 17. PMID 37847518

RESULTS

PARTICIPANT FLOW:
Groups:
- Third Dose BNT162b2: This group received BNT162b2 (Pfizer-BioNTech) as their third dose.
- Third Dose mRNA-1273: This group received mRNA-1273 (Moderna) as their third dose
Period: Overall Study
Arm/Group | Third Dose BNT162b2 | Third Dose mRNA-1273
Started | 137 | 136
Completed | 119 | 125
Not Completed | 18 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Third Dose BNT162b2 | Third Dose mRNA-1273 | Total
Number analyzed (Participants) | 137 | 136 | 273
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71 [61 to 79] | 69 [57 to 77] | 70 [59 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 57 | 121
  Male | 73 | 79 | 152
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 66 | 67 | 133
  Black or African origin | 10 | 13 | 23
  White | 33 | 29 | 62
  Other/multiracial | 18 | 17 | 35
  Missing | 10 | 10 | 20
Baseline two dose COVID-19 vaccine type [Count of Participants; unit: Participants]
  mRNA-1273 | 56 | 55 | 111
  BNT162b2 | 81 | 81 | 162
Days between COVID-19 vaccine doses, median [Median (Inter-Quartile Range); unit: Days]
  First and second dose | 28 [25 to 35] | 28 [28 to 33] | 28 [27 to 35]
  Second dose and third dose | 253 [203 to 306] | 252 [215 to 306] | 252 [206 to 306]
eGFR category [Count of Participants; unit: Participants]
  30-44 ml/min per 1.73 m2 | 5 | 4 | 9
  15-29 ml/min per 1.73 m2 | 1 | 2 | 3
  <15 ml/min per 1.73 m2 (nondialysis) | 2 | 2 | 4
  Dialysis | 129 | 128 | 257
Nondialysis CKD participants - eGFR by CKD-EPI [Median (Inter-Quartile Range); unit: ml/min per 1.73 m2] — Population: Non-dialysis CKD participants only
  ml/min per 1.73 m2
    number analyzed (Participants) | 8 | 8 | 16
    (all) | 33 [23 to 37] | 31 [24 to 33] | 31 [24 to 35]
Nondialysis CKD participants - Microalbumin to creatinine ratio [Mean (Standard Deviation); unit: mg/mmol] — Population: Nondialysis CKD participants only
  mg/mmol
    number analyzed (Participants) | 8 | 8 | 16
    (all) | 531 (692) | 725 (800) | 628 (729)
Dialysis modality [Count of Participants; unit: Participants] — Population: Only applicable to dialysis patients
  Participants
    In-center hemodialysis: number analyzed (Participants) | 129 | 128 | 257
    In-center hemodialysis | 122 | 119 | 241
    Home hemodialysis: number analyzed (Participants) | 129 | 128 | 257
    Home hemodialysis | 5 | 5 | 10
    PD: number analyzed (Participants) | 129 | 128 | 257
    PD | 2 | 4 | 6
Dialysis access [Count of Participants; unit: Participants] — Population: Only applicable for Dialysis patients
  Participants
    Central venous catheter: number analyzed (Participants) | 129 | 128 | 257
    Central venous catheter | 78 | 76 | 154
    Arteriovenous fistula or graft: number analyzed (Participants) | 129 | 128 | 257
    Arteriovenous fistula or graft | 49 | 48 | 97
    PD catheter: number analyzed (Participants) | 129 | 128 | 257
    PD catheter | 2 | 4 | 6
Dialysis vintage [Median (Inter-Quartile Range); unit: years] — Population: For dialysis patients only
  years
    number analyzed (Participants) | 129 | 128 | 257
    (all) | 2.6 [1.5 to 4.6] | 2.6 [1.5 to 4.6] | 2.6 [1.3 to 4.7]
Cause of kidney disease [Count of Participants; unit: Participants]
  Ischemic nephropathy | 34 | 25 | 59
  Diabetes mellitus | 63 | 63 | 126
  Glomerulonephritis | 20 | 26 | 46
  Cystic kidney disease | 3 | 7 | 10
  Other/unknown | 17 | 15 | 32
Prior COVID-19 infection [Count of Participants; unit: Participants]
  COVID-19 (RT-PCR confirmed) | 5 | 3 | 8
  Symptomatic COVID-19 | 2 | 3 | 5
  COVID-19 hospitalization | 2 | 1 | 3
  COVID-19 intensive care unit admission | 1 | 1 | 2
Comorbidities [Count of Participants; unit: Participants]
  Active smoker | 7 | 5 | 12
  Chemotherapy (3 mo) | 3 | 2 | 5
  Chronic obstructive lung disease | 5 | 10 | 15
  Coronary artery disease | 12 | 19 | 31
  Congestive heart failure | 24 | 17 | 41
  Cerebrovascular disease | 8 | 7 | 15
  Hepatitis B nonresponder (HbsAb ,10 mIU/ml) | 52 | 58 | 110
  Hypertension | 118 | 112 | 230
  Immunosuppression | 3 | 4 | 7
  Malignancy (prior 5 yr) | 9 | 9 | 18
  Myocardial infarction | 17 | 8 | 25
  Obesity (BMI $30 kg/m2) | 13 | 15 | 28
  Peripheral vascular disease | 13 | 7 | 20
  Solid organ transplant | 27 | 19 | 46
  Type 1 diabetes mellitus | 6 | 5 | 11
  Type 2 diabetes mellitus | 84 | 72 | 156

OUTCOME MEASURES:

1. Primary Outcome: Serum Level of Anti-RBD ( Anti Receptor Binding Domain )
Description: To measure Anti-Spike, Anti-NP antibodies, and SARS-CoV-2 specific neutralization at 1 month (30 days) following third dose of vaccine (BNT162b2 versus mRNA-1273) binding antibody levels for anti-receptor-binding domain and antispike IgG were reported as relative ratios to a synthetic standard included as a calibration curve on each assay plate.
Time Frame: One month
Population: 7 participants withdrew from each arm and were not included in analysis. Only participants who provided samples for this timepoint were included in the analysis.
Measure: Mean (Standard Deviation); unit: relative ratio
Arm/Group | Third Dose BNT162b2 | Third Dose mRNA-1273
Number analyzed (Participants) | 126 | 125
relative ratio
  Anti-NP | 0.0630 (0.334) | 0.0415 (0.169)
  Anti-RBD | 0.807 (0.416) | 0.934 (0.398)
  Anti-spike | 1.26 (0.358) | 1.33 (0.289)

2. Secondary Outcome: Serum Level of SARS-CoV-2 Antibodies
Description: To determine the effect of a third dose of COVID-19 vaccine on humoral immune response in hemodialysis patients through measurement of Anti-Spike, Anti-RBD, and Anti-NP antibodies at 3 months binding antibody levels for anti-receptor-binding domain and antispike IgG were reported as relative ratios to a synthetic standard included as a calibration curve on each assay plate.
Time Frame: 3 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: relative ratios
Arm/Group | Third Dose BNT162b2 | Third Dose mRNA-1273
Number analyzed (Participants) | 119 | 121
relative ratios
  Anti-NP | 0.0985 (0.424) | 0.0665 (0.178)
  Anti-RBD | 0.787 (0.479) | 0.941 (0.499)
  Anit-Spike | 1.14 (0.389) | 1.24 (0.360)

3. Secondary Outcome: Serum Level of SARS-CoV-2 Antibodies
Description: To determine the effect of a third dose of COVID-19 vaccine on humoral immune response in hemodialysis patients through measurement of Anti-Spike, Anti-RBD, and Anti-NP antibodies at 6 months binding antibody levels for anti-receptor-binding domain and antispike IgG were reported as relative ratios to a synthetic standard included as a calibration curve on each assay plate.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: relative ratios
Arm/Group | Third Dose BNT162b2 | Third Dose mRNA-1273
Number analyzed (Participants) | 28 | 29
relative ratios
  Anti-NP | 0.0703 (0.173) | 0.0711 (0.132)
  Anti-RBD | 0.658 (0.438) | 0.819 (0.463)
  Anti-Spike | 1.16 (0.403) | 1.30 (0.302)

4. Secondary Outcome: Serum Level of SARS-CoV-2 Antibodies
Description: Determine the effect of a third dose of COVID-19 vaccine on humoral immune response in hemodialysis patients through measurement of Anti-Spike, Anti-RBD, and Anti-NP antibodies at 12 months
Time Frame: 12 months
Population: Study was terminated before 12 months visit occurred.
Arm/Group | Third Dose BNT162b2 | Third Dose mRNA-1273
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Proportion of B and T-cell Lymphocyte Subsets in Peripheral Blood Mononuclear Cells (PBMC)
Description: In a subset of participants, assess cellular immunity through flow cytometry on PBMC and single-cell RNA sequencing prior to, one month, and 6 months following vaccine booster.
Time Frame: 1 month
Population: Analysis on this subset was not feasible following study completion. The collaborating laboratory was unable to logistically perform this testing due to the resources required for Flow Cytometry, and therefore this secondary outcome was not analyzed.
Arm/Group | Third Dose BNT162b2 | Third Dose mRNA-1273
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Adverse Event
Description: Evaluate adverse events related to third dose of vaccine through a questionnaire within 48 hours to 14 days following third vaccine dose.
Time Frame: 14 days
Population: Population consists of only individuals who returned the completed survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Third Dose BNT162b2 | Third Dose mRNA-1273
Number analyzed (Participants) | 129 | 126
Participants
  Pain | 67 | 76
  Redness | 2 | 6
  Swelling | 2 | 9
  Fever (38°C) | 4 | 14
  Chills | 8 | 19
  Fatigue | 17 | 30
  Nausea or vomiting | 6 | 10
  Diarrhea | 2 | 2
  Myalgia | 15 | 13
  Arthralgia | 2 | 5
  Headache | 12 | 15
  Any symptom | 82 | 89
  Any severe symptom | 10 | 12
  Any systemic symptom | 36 | 55
  Antipyretic medication | 29 | 42

7. Secondary Outcome: Adverse Events (30 Days)
Description: Evaluate adverse events related to third dose of vaccine through a questionnaire at 30 days following third vaccine dose.
Time Frame: 1 month
Population: We did not systematically collect symptoms at 30 days following vaccine dose, but rather 2-14 days only. This outcome was not analyzed.
Arm/Group | Third Dose BNT162b2 | Third Dose mRNA-1273
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Hospitalization
Description: Number of participants who experienced COVID-19 related hospitalizations by study groups.
Time Frame: 6 months
Population: 7 participants withdrew from each arm
Measure: Count of Participants; unit: Participants
Arm/Group | Third Dose BNT162b2 | Third Dose mRNA-1273
Number analyzed (Participants) | 130 | 129
Participants | 1 | 2

9. Secondary Outcome: COVID-19 Infections
Description: Number of participants who experienced COVID-19 infections and symptomatic COVID-19 infections.
Time Frame: 6 months
Population: 7 participants withdrew from each arm
Measure: Count of Participants; unit: Participants
Arm/Group | Third Dose BNT162b2 | Third Dose mRNA-1273
Number analyzed (Participants) | 130 | 129
Participants
  Confirmed cases of COVID-19 Infections | 11 | 15
  Confirmed cases of COVID-19 Infections with symptoms: number analyzed (Participants) | 11 | 15
  Confirmed cases of COVID-19 Infections with symptoms | 3 | 10

10. Secondary Outcome: Death
Description: Differences in death between study groups. Death was collected for 6 months following third dose (shorted from 12 months due to the introduction of the 4th dose).
Time Frame: 6 months
Population: excludes 7 participants that withdrew from each arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Third Dose BNT162b2 | Third Dose mRNA-1273
Number analyzed (Participants) | 130 | 129
Participants | 17 | 9

ADVERSE EVENTS:
Time Frame: Deaths and serious adverse events were assessed for 6 months following 3rd dose and vaccine related (non-serious) adverse events were assessed over 2-14 days post-third dose.
Description: All participants dosed were assessed for Deaths and Serious Adverse Events through self-report/review of EMR.
  Other (non-serious) adverse events were systematically collected 2-14 days post third dose from participants who returned a questionnaire (129 from BNT162b2 and 126 from mRNA-1273).
Arm/Group | Third Dose BNT162b2 | Third Dose mRNA-1273
All-Cause Mortality (participants affected / at risk) | 17/137 | 9/136
Serious Adverse Events (participants affected / at risk) | 23/137 | 16/136
Other Adverse Events (participants affected / at risk) | 82/129 | 89/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Third Dose BNT162b2 (N=137) | Third Dose mRNA-1273 (N=136)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Axillary abscess (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cardiac arrest (Cardiac disorders) | 4 (4) | 2 (2)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Colitis / Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death, unspecified (General disorders) | 3 (3) | 2 (2)
End stage renal disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Hypervolaemia (Cardiac disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Ischaemic stroke (Vascular disorders) | 1 (1) | 0 (0)
Multiple myeloma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Mycotic pseudoaneurysm of aorta (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0 (0)
Anema (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Cerebral Infarction (Vascular disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Myocardial infarction (Vascular disorders) | 0 (0) | 1 (1)
Peripheral swelling (Cardiac disorders) | 0 (0) | 1 (1)
Seizures (Nervous system disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 3 (3)
Steal phenomenon (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Third Dose BNT162b2 (N=129) | Third Dose mRNA-1273 (N=126)
Pain (Skin and subcutaneous tissue disorders) | 67 (67) | 76 (76) — Local injection site reaction - Pain
Redness (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (6) — Local injection site reaction - Redness
Swelling (Skin and subcutaneous tissue disorders) | 2 (2) | 9 (9) — Local injection site reaction - Swelling
Fever (38 degrees) (Immune system disorders) | 4 (4) | 14 (14)
Chills (Immune system disorders) | 8 (8) | 19 (19)
Fatigue (Immune system disorders) | 17 (17) | 30 (30)
Nausea of vomiting (Gastrointestinal disorders) | 6 (6) | 10 (10)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 15 (15) | 13 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (5)
Headache (Nervous system disorders) | 12 (12) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-05): https://cdn.clinicaltrials.gov/large-docs/29/NCT05022329/Prot_SAP_000.pdf